CLINICAL TRIAL: NCT06669962
Title: Characterisation of the Biochemical Profile and Physiology of the Coronary Circulation in Takotsubo Syndrome
Acronym: TAKO-PROVE
Status: Recruiting | Type: Observational
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Sponsor
Other Study IDs: AOUCitta
Record Dates: First submitted 2024-07-04; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-07

CONDITIONS: Tako Tsubo Cardiomyopathy
MeSH Terms: conditions — Takotsubo Cardiomyopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — peripheral blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Study of coronary microcirculation and biomarkers of microvascular dysfunction — Patients with tako-tsubo syndrome will undergo to coronary angiography, ventriculography and assessment of physiological indexes of coronary circulation as per clinical practice

SUMMARY:
Consecutive consenting patients over the age of 18 years diagnosed with Takotsubo syndrome according to the position statement of the European Journal of Heart Failure (2016) will be included in the study. The primary endpoint is to evaluate the incidence of coronary microcirculation dysfunction and its correlation with the clinical presentation and the prognosis in patients with TAKO-Tsubo syndrome. Secondary endpoints will be to assess the incidence of in-hospital mortality, the prevalence of cardiogenic shock, the correlation between the levels of biomarkers analyzed, microvascular dysfunction, perceived quality of life, and angina severity during hospitalization and at subsequent follow-ups, and the influence of knowledge of the level of microvascular dysfunction on clinical management and prescribed therapies. Enrolment: 2 years, follow-up: 1 month and 1 year. Total: 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Diagnosis of Takotsubo syndrome
* Signing of informed consent

Exclusion Criteria:

* Age <18 years;
* Refusal to sign written informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive consenting patients over the age of 18 years with a diagnosis of Takotsubo syndrome will be included in the study according to the position statement of the European Journal of Heart Failure (2016).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2026-06-27 (Estimated); Study Completion 2027-06-27 (Estimated)

PRIMARY OUTCOMES:
Incidence of coronary microcirculation dysfunction | one year
  coronary microvascular dysfunztion will be defined as a coronary flow reserve (CFR) < 2.5 and/or as an index of microvascular resistance (IMR) > 25 , as assessed with Coroventis syestem

SECONDARY OUTCOMES:
Incidence of in-hospital mortality | up to thirty days
  all-cause death
Correlation between the levels of biomarkers analysed and microvascular dysfunction | at discharge (assessed up to 5 days)
  Several biomarkers (namely neuropeptide Y, troponin I, nt-pro BNP) will be measured via center-specific labratory essays) and a correlation of their blood levels with coronary microvascular dysfunction ( coronary flow reserve (CFR) and index of microvascular resistance (IMR) assessed with Coroventis system) will be sought
Perceived quality of life | one year
  Assessed with Euro Quality of life scale 5D (EQOL-5d): EQ-5D descriptive system is a preference-based HRQL measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort,and anxiety/depression. The answers given to ED-5D permitto find 243 unique health states or can be converted into EQ-5D index an utility scores anchored at 0 for death and 1 for perfect health. The EQ-5D questionnaire also includes a Visual Analog Scale (VAS), by which respondents can report their perceived health status with a grade ranging from 0 (the worst possible health status) to 100 (the best possiblehealth status).
Severity of angina | one year
  assessed with the Seattle Angina Questionnaire (SAQ): This SAQ quantifies 5 domains measuring the impact of angina on patients' health status: Physical Limitation (9 items), Angina Stability (1item), Angina Frequency (2 items), Treatment Satisfaction (4 items), and Quality of Life (3 items). Item responses are coded sequentially from worst to best status and range from 1 to 6 for Physical Limitation, Angina Stability, and Angina Frequency items; 1 to 5/6 for Treatment Satisfaction items; and 1 to 5 for Quality of Life items

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Città della Salute e della Scienza, Turin, Turin, Italy

IPD SHARING:
Plan to Share IPD: No